CLINICAL TRIAL: NCT04809506
Title: Bio-collection for the Discovery of New Biomarkers for the Prediction of Cardiovascular Events
Brief Title: Identification of New Biomarkers for the Prediction of Cardiovascular Events
Acronym: CDPA-Biobank
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0116
Record Dates: First submitted 2021-03-11; First posted 2021-03-22 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases
Keywords: Arterial disease; atherosclerosis; Thrombosis; Biomarkers; Genetic polymorphisms
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient consulting the Centre for Screening and Prevention of Atherosclerosis: 2 additional blood samples (2 x 7ml) at every visit
  Interventions: Biological: additional blood samples

INTERVENTIONS:
Biological: additional blood samples — 2 additional blood samples (2 x 7ml) at every visit

SUMMARY:
The main goal of this project is to constitute a collection of biological samples, obtained through the clinical activity of the Centre for Screening and Prevention of Atherosclerosis at Toulouse University Hospital, managing patients in primary or secondary prevention for cardiovascular (CV) diseases. The main objective is to validate new biomarkers with prognostic value regarding the onset of future CV events. Besides, the biological collection will enable patho-physiological studies on atherosclerosis related diseases.

DETAILED DESCRIPTION:
Cardiovascular (CV) diseases, particularly those secondary to atherosclerosis, are a leading cause of morbidity and mortality in modern societies. Classical CV risk factors, including age and gender, family history, tobacco smoking, hypertension, diabetes, dyslipidemia and obesity cannot predict more than 50% of future CV events. Use of specific scores (like the SCORE chart) does not much contribute to the precise evaluation of patients classified at moderate risk. Thus, more research is needed: 1) to study patho-physiological mechanisms of the atherothrombotic process in order to identify new pharmacological targets and, 2) to validate new biomarkers with a strong predictive value regarding the onset of hard CV clinical events. Moreover, genetic polymorphisms underlie an individual's susceptibility to develop atherosclerotic diseases. Identification of those gene variants might help to define a personalized approach for the treatment of CV diseases. Patients consulting the Centre for Screening and Prevention of Atherosclerosis (CDPA) are submitted to a personal face-to-face interview addressing their life style, nutritional and smoking habits, and their physical activity practice. Clinical examination includes ECG, stress test, ankle-arm systolic index, ultrasonography of arteries (carotid, aorta, lower limb) and determination of a coronary calcification score. Blood samples are taken up for chemistry measurements including lipoproteins (triglycerides, LDL-C, HDL-C, Lp(a)). For the specific purpose of the biological collection, two supplementary blood tubes will be collected (2 x 7 ml); serum, plasma and genomic DNA will be prepared. Patients will be followed up yearly for those on secondary prevention and every 2nd year on primary prevention. Identical investigation will be carried out at every visit. Recruitment period will spread over 5 years and follow-up will be pursued up to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 yrs;
* consulting the Centre for Screening and Prevention of Atherosclerosis (CDPA) for management of their cardiovascular risk factors;
* patients on primary prevention, free of personal history of coronary artery disease, stroke or lower limb arteriopathy, or patients on secondary prevention having presented one of the above mentioned diseases;
* patients affiliated to a health insurance system;
* patients having given their written informed consent for a participation to the study and for possible genetic analysis of their personal traits.

Exclusion Criteria:

* Patients under the age of 18;
* patients being under legal protection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting the Centre for Screening and Prevention of Atherosclerosis (CDPA) for management of their cardiovascular risk factors; patients on primary prevention, free of personal history of coronary artery disease, stroke or lower limb arteriopathy, or patients on secondary prevention having presented one of the above mentioned diseases
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2030-02-03 (Estimated); Study Completion 2034-02-03 (Estimated)

PRIMARY OUTCOMES:
measurement of the candidate biomarker | Day 0
  measurement, at baseline of the candidate biomarker, with respect to the onset, during follow-up, of a cardiovascular event: either coronary events or cerebrovascular stroke or lower limb arteriopathy.
measurement of the candidate biomarker | during the intervention/procedure/surgery
  measurement, at baseline of the candidate biomarker, with respect to the onset, during follow-up, of a cardiovascular event: either coronary events or cerebrovascular stroke or lower limb arteriopathy.

SECONDARY OUTCOMES:
evolution of clinical and biological parameters involved in atherothrombosis | Day 0
  Pathophysiological mechanisms involved in atherothrombosis will be investigated using biomarkers addressing specific pathways: lipid metabolism, inflammation, endothelial reactivity, myocardial function. For a given new biomarker, its transferability to a clinical lab will be evaluated by its analytical performances and its possible adaptation to a semi-automated platform.
evolution of clinical and biological parameters involved in atherothrombosis | during the intervention/procedure/surgery
  Pathophysiological mechanisms involved in atherothrombosis will be investigated using biomarkers addressing specific pathways: lipid metabolism, inflammation, endothelial reactivity, myocardial function. For a given new biomarker, its transferability to a clinical lab will be evaluated by its analytical performances and its possible adaptation to a semi-automated platform.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Ferrieres, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No